CLINICAL TRIAL: NCT03445871
Title: Association Between Methotrexate Erythrocyte Polyglutamate Concentration and Clinical Response in Rheumatoid Arthritis Patients Treated With Subcutaneous Injectable Methotrexate
Acronym: POLYGLU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1708155; 2017-004348-39 (EudraCT Number)
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Methotrexate; Erythrocyte polyglutamate; Compliance Questionnaire Rheumatology
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with active rheumatoid arthritis (Active Comparator): Patients with active rheumatoid arthritis will be included. They will have a blood sample and Compliance Rheumatology Questionnaire (CRQ).
  Interventions: Biological: Blood sample; Diagnostic Test: CRQ
- Patients with rheumatoid arthritis into remission (Active Comparator): Patients with rheumatoid arthritis into remission will be included. They will have a blood sample and Compliance Rheumatology Questionnaire (CRQ).
  Interventions: Biological: Blood sample; Diagnostic Test: CRQ

INTERVENTIONS:
Biological: Blood sample — Blood samples will be collected for measuring PG-MTX blood concentration.
Diagnostic Test: CRQ — Compliance Rheumatology Questionnaire (CQR) is a self-administered questionnaire for to evaluate therapeutic observance during rheumatoid arthritis.
  Other Names: Compliance Rheumatology Questionnaire

SUMMARY:
Methotrexate (MTX) is the first-line treatment of rheumatoid arthritis (RA). In case of MTX failure, it is discussed to start a Biologic Disease-modifying Antirheumatic Drug (bDMARDs) according to the latest European recommendations of the EULAR. Before to add a Biologic Disease-modifying Antirheumatic Drug (bDMARDs), an objective estimation of MTX impregnation could be carried out by MTX polyglutamates (MTX-PG). In rheumatoid arthritis patients with active disease estimated by DAS28 (Disease activity Score 28)> 3.2 insufficiently controlled by MTX subcutaneously and patients in remission obtained with a DAS 28 <2.6 with methotrexate prescribed since more than 6 months at stable dose for at least 3 months, a concentration of MTX-PG will be achieved.

DETAILED DESCRIPTION:
The assumption is the association between low methotrexate erythrocyte polyglutamate and low clinical response in rheumatoid arthritis patients treated with subcutaneous injectable methotrexate. Adherence to MTX will be assessed by the Compliance Questionnaire Rheumatology (CQR). Measurement of this adherence could optimize MTX treatment prior to the use of biotherapy which is costly with a lower infectious tolerance.

Correlation between its concentration and compliance assessed by CQR questionnaire will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and have social security affiliation.
* Patients followed in the Rheumatology Department at the hospital of St Etienne.
* Patients with rheumatoid arthritis and :

  * Either Rheumatoid arthritis patients in remission (DAS 28<2.6) with MTX treatment for at least 6months, and with a stable dose for 3months.
  * Or patients with a High Disease Activity Rheumatoid Arthritis activity (DAS 28>3.2) with MTX treatment (≥ 15 mg/weeks), taking MTX treatment for at least 6months with a stable subcutaneous weekly MTX injection (≥ 15 mg/weeks) treatment during the previous 3 months.
* Signed informed consent.

Exclusion Criteria:

* Patients treated with another conventional synthetic Disease Modifying Anti-Rheumatic Drugs (csDMARD)
* Another diagnostic than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
MTX-PG concentration | Hour 1
  To compare MTX-PG concentration in patients with active rheumatoid arthritis and patients with rheumatoid arthritis in remission

SECONDARY OUTCOMES:
different metabolites dosing of MTX-PG | Hour 1
  Analysis of different metabolites dosing of MTX-PG by High-performance liquid chromatography technical
CQR score | Hour 1
  Analysis of CQR score response

CONTACTS AND LOCATIONS:
Overall Officials: Hubert MAROTTE, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No